CLINICAL TRIAL: NCT05789316
Title: Head and Neck Cancer Survivorship Ototoxicity Screening (SOS) Protocol
Brief Title: Head and Neck Cancer Survivorship Ototoxicity Screening (SOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202302038
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer Survivors; Cancer of the Head and Neck Surviors
Keywords: survivorship; quality of life; cisplatin; radiation; head and neck cancer; hearing loss; ototoxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Hearing Loss; Ototoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ototoxicity Screening Protocol (Experimental): After enrollment, participants will complete a pre-screening survey. Before their survivorship clinic visit, participants will complete the ototoxicity screening protocol and implementation outcome surveys. During their visit, they will receive counseling on ototoxicity and referral to audiology. After their visit, they will complete the SESMQ and WU-QOLv4 surveys and undergo pure tone audiometry. Each participant will complete this protocol once. The investigators will follow each participant by chart review for at least six months to evaluate for audiologic follow-up.
  Interventions: Other: Ototoxicity Screening Protocol

INTERVENTIONS:
Other: Ototoxicity Screening Protocol — The ototoxicity screening protocol contains a functional and objective component. The functional component is the Hearing Handicap Inventory for the Elderly - Screening Version (HHIE-S). The objective component will be pure tone audiometry. A 2 kHz tone at 40 dB will play through over-the-ear headphones and subjects will indicate whether they heard it.

SUMMARY:
To evaluate the effectiveness, feasibility, acceptability, and appropriateness of an ototoxicity screening protocol among head and neck (H&N) cancer patients followed in survivorship clinic that received cisplatin-based chemoradiation therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old)
* H&N cancer patients will be eligible for inclusion if they have previously undergone cisplatin-based CRT or radiotherapy, including proton therapy, intensity-modulated radiation therapy, and adaptive radiotherapy-surgery with curative intent (i.e., definitive, neoadjuvant, or adjuvant) or definitive surgery with neoadjuvant or adjuvant radiation.

Exclusion Criteria:

* Patient has been evaluated by an audiologist within the past 12 months
* Use of a hearing aid
* Received a cochlear implant
* Cannot complete simple forms in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Rate of participants who complete audiologic follow-up | Through completion of follow-up (estimated to be 6 months)

SECONDARY OUTCOMES:
Feasibility of ototoxicity screening protocol as measured by the Feasibility of Intervention Measure | Before survivorship clinic visit (Day 1)
  -Contains 4 statements about the proposed intervention that are scored on a five-point Likert scale (1 indicates the participant "completely disagrees", 5 indicates "completely agrees"). A score greater than or equal to 4 will indicate the intervention is feasible.
Acceptability of ototoxicity screening protocol as measured by the Acceptability of Intervention Measure | Before survivorship clinic visit (Day 1)
  -Contains 4 statements about the proposed intervention that are scored on a five-point Likert scale (1 indicates the participant "completely disagrees", 5 indicates "completely agrees"). A score greater than or equal to 4 will indicate the intervention is acceptable.
Appropriateness of ototoxicity screening protocol as measured by the Intervention Appropriateness Measure | Before survivorship clinic visit (Day 1)
  -Contains 4 statements about the proposed intervention that are scored on a five-point Likert scale (1 indicates the participant "completely disagrees", 5 indicates "completely agrees"). A score greater than or equal to 4 will indicate the intervention is appropriate.
Functional hearing loss of participants as measured by the Situational Management Questionnaire (SESMQ) | After survivorship clinic visit (Day 1)
  -This questionnaire contains 20 situations. Participants rate each situation according to their ability to hear in the given situation (hearing ability scale; SESMQH) and their confidence in managing the given situation (confidence scale; SESMQC). The score for each situation ranges from 0 (poor hearing/low confidence) to 10 (normal hearing/high confidence), totaling 200 points for each scale. The higher the score indicates less hearing loss to the participant.
Quality of life of participants as measured by the University of Washington Quality of Life Questionnaire (UW-QOL) | After survivorship clinic visit (Day 1)
  -This questionnaire contains 16 items on morbidities associated with H&N cancer treatment. Twelve items are graded on a 5-point Likert scale. One question lists treatment-related morbidities and ask participants to identify their top three most important issues. The last three questions evaluate global QoL. It is scored on a scale from 0 (worst) to 100 (best). However, UW-QOL does not include symptoms of ototoxicity. Therefore, the investigators will modify it to include tinnitus and hearing loss as additional 5-point Likert scale questions and morbidities in the rank order question.
Functional social support as measured by the Duke-UNC Functional Social Support Questionnaire | After survivorship clinic visit (Day 1)
  It has been validated for use in populations of cancer patients and cancer survivors. 5 questions are presented using a Likert scale from 0-2, with higher scores indicating a higher level of social support.

CONTACTS AND LOCATIONS:
Overall Officials: David Lee, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu